CLINICAL TRIAL: NCT02227797
Title: MT2013-37R: Voriconazole Therapeutic Drug Monitoring in Pediatric Hematopoietic Stem Cell Transplant Patients
Brief Title: MT2013-37R: Voriconazole Monitoring in Pediatric Stem Cell Transplant Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013LS126; MT2013-37R
Record Dates: First submitted 2014-08-26; First posted 2014-08-28 (Estimated); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Fungal Infection
Keywords: stem cell transplant; hematopoietic stem cell transplant; fungal infection; voriconazole; pediatric
MeSH Terms: conditions — Mycoses | interventions — Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Voriconazole (Experimental)
  Interventions: Drug: Voriconazole

INTERVENTIONS:
Drug: Voriconazole — 6 mg/kg to 12 mg/kg IV/PO every 12 hours depending on patient age and dose toleration of prior patients

SUMMARY:
The primary purpose of this study is to identify the optimal dose of voriconazole, an anti-fungal drug often used in people undergoing stem cell transplant. An optimal dose level is one level that provides a good blood level (concentration) of voriconazole without too much toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing allogeneic hematopoietic stem cell transplantation (either 1st or subsequent)
* Age ≤ 21 years
* Adequate organ function within 14 days of enrollment, i.e. Creatinine: < 1.5 x ULN and Hepatic: ALT, AST and total bilirubin < 3 x ULN
* Requires voriconazole to prevent or treat invasive fungal infection after undergoing stem cell transplantation

Exclusion Criteria:

* Has received voriconazole within 5 days prior to starting study therapy
* History of hypersensitivity or severe intolerance to azoles
* History, or current evidence, of cardiac arrhythmias defined as QTc ≥ 480 mm/sec
* Receiving the following drugs and cannot be discontinued at least 24 hours before starting therapy: pimozide, quinidine, astemizole, ergot alkaloids.
* Received one or more of the following drugs within 14 days prior to starting study, as they are potent inducers of hepatic microsomal enzymes: rifampin, rifabutin, carbamazepine, phenytoin, nevirapine, long-acting barbiturates.
* Received sirolimus within the 14 days prior to starting study as voriconazole is a potent inhibitor of sirolimus metabolism
* Receiving or anticipated need for methadone as co-administration with voriconazole potentially increases methadone exposure

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Actual)
Dates: Start 2015-01-19 (Actual); Primary Completion 2017-09-08 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated, minimum efficacious dose for 3 different pediatric age groups | Seven days after starting voriconazole

SECONDARY OUTCOMES:
Correlation of initial dose of voriconazole with voriconazole blood concentration in 3 different pediatric age groups | After starting voriconazole: Day 5, between Days 12-15, between Days 19-22
Correlation of voriconazole dose with elevations to 5 times the upper limit of normal in liver enzymes | After starting voriconazole: Twice a week Days 1-30 and 1 week after the last dose of voriconazole ~ Day 35-42
Incidence of fungal infection | 6-month period after transplant

CONTACTS AND LOCATIONS:
Overall Officials: Angela Smith, M.D., Principal Investigator — Masonic Cancer Center, University of Minnesota; Pui-Yang Iroh Tam, M.D., Principal Investigator — Masonic Cancer Center, Univeristy of Minnesota
Locations (1):
- University of Minnesota Medical Center, Fairview, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Takahashi T, Jaber MM, Smith AR, Jacobson PA, Fisher J, Kirstein MN. Predictive Value of C-Reactive Protein and Albumin for Temporal Within-Individual Pharmacokinetic Variability of Voriconazole in Pediatric Patients Undergoing Hematopoietic Cell Transplantation. J Clin Pharmacol. 2022 Jul;62(7):855-862. doi: 10.1002/jcph.2024. Epub 2022 Feb 19. PMID 34970774